CLINICAL TRIAL: NCT03883438
Title: Coronally Advanced Flap and Envelope Type of Flap Plus Acellular Dermal Matrix Graft for the Treatment of Thin Phenotype Multiple Recession Defects
Brief Title: Cor Adv Flap Plus Ac Derm Matrix in Thin Phenotype Multiple Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aziz Aliyev Azerbaijan State Advanced Training Institute for Doctors (Other)
Collaborators: Altinbas University (Other); Universidade Ibirapuera (Other); Universidad El Bosque, Bogotá (Other)
Responsible Party: Principal Investigator, Cavid Ahmedbeyli, Associate Professor, Aziz Aliyev Azerbaijan State Advanced Training Institute for Doctors
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AZETR201520171001
Record Dates: First submitted 2019-03-17; First posted 2019-03-20 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Gingival Recession, Generalized
Keywords: Gingival recession; Therapy; Surgery; Tooth root; Surgical flaps; Acellular dermis
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: A total of 22 patients with 55 recessions were included in this single blind randomized controlled trial. Each patient had at least two recessions with a depth of ≥ 3 mm (Miller Class I&II) in the upper jaw. The entry criteria were esthetic indication for root coverage; absence of caries or restorations at the selected sites; no history of previous mucogingival therapy; being a non-smoker and a systemically healthy patient.
Who Masked: Participant
Masking Description: A computer program was used to randomize 22 volunteers to treatment groups by a person who was not involved in the study. The result of this randomization process was written on a paper and then put in the sealed opaque envelope by a blinded examiner, in which the treatment procedure for the specific patient was defined. The envelope was opened by surgeon, immediately before starting the surgical procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coronally advanced flap and acellular dermal graft (Active Comparator): In CAF group, after local anesthesia oblique beveled vertical incisions were made at the most mesial and distal line angles of the recessions. These two incisions were connected with an intra-sulcular and interdental sub-marginal incisions in order to create the external surgical papillae. Then the flap was elevated as a split-full-split approach. The apical portion of the flap was reflected as close to the periosteum as possible by mesio-distal and apical sharp dissection parallel to the mucosa to release residual muscle tension and extended beyond the muco-gingival junction to facilitate the passive coronal replacement of the flap over the defects. In both groups ADMG was used as a sub-epithelial graft considering the manufacturer's instructions. The graft was positioned at the level of cemento-enamel junction and extended to the surrounding bone in the apical direction with full closure of the exposed root surfaces.
  Interventions: Procedure: Modified coronally advanced flap and acellular dermal matrix graft
- Modified coronally advanced flap and acellular dermal graft (Experimental): Test group received CAF avoiding vertical releasing incisions (mCAF).
  Interventions: Procedure: Modified coronally advanced flap and acellular dermal matrix graft

INTERVENTIONS:
Procedure: Modified coronally advanced flap and acellular dermal matrix graft — Evaluation of the effectiveness of vertical incisions in the management of multiple gingival recessions (Miller Class I&II ≥3 mm) treated with coronally advanced flap and acellular dermal matrix graft

SUMMARY:
Clinical evaluation of conventional and modified coronally advanced flaps combined with acellular dermal matrix graft

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effectiveness of vertical incisions in the management of multiple gingival recessions (Miller Class I&II ≥3 mm) treated with coronally advanced flap (CAF) and acellular dermal matrix graft (ADMG) in 22 eligible participants.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients
* Miller Class I & II multiple buccal recession defects ≥ 3 mm on maxillary incisors, canines or premolars
* Esthetic indication for root coverage
* Probing depth < 3mm at the recession sites

Exclusion Criteria:

* Smokers
* Pregnancy
* Bruxism and occlusal trauma
* Previous root coverage procedure
* Endodontically treated teeth at the recession sites
* Caries or restorations at the recession sites
* Use of antibiotics over the previous 3 months prior to treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-02-15 (Actual)

PRIMARY OUTCOMES:
Complete root coverage | 12 months
  Complete defect coverage was calculated as the percentage of patients with defects having complete coverage achieved as the gingival margin at cemento-enamel junction or coronal level.
Root coverage esthetic score | 12 months
  Root coverage esthetic score (RES) was used as a scoring system to assess the esthetic outcomes following root coverage procedures on Miller Class I & II gingival recession defects through the evaluation of clinical cases. Gingival margin level, marginal tissue contour, soft tissue texture, mucogingival junction alignment and gingival color were evaluated without magnification. Zero, 3 and 6 points were used for the evaluation of the position of the gingival margin, whereas a score 0 or 1 point was used for each of the other variables.
Patient satisfaction score | 12 months
  Each patient was questioned about his/her satisfaction with regard to the following patient-centered criteria:
  Root coverage attained, relief from dentinal hypersensitivity, color of gums, shape and contour of gums, surgical procedure in terms of pain during surgery and the discomfort experienced related to the duration of the procedure and handling by the operator, post surgical phase in terms of the pain, swelling, and postoperative complications; and cost effectiveness in terms of the time and money spent for the treatment.
  Patient satisfaction was assessed using a three-point rating scale: fully satisfied (3 points); satisfied (2 points); and unsatisfied (1 point).

SECONDARY OUTCOMES:
Plaque Index | 12 months
  Teeth were isolated by cotton rolls and after drying by air syringe, the microbial dental plaque was evaluated by the explorer from 4 tooth surfaces (mesio-buccal, mid-buccal, disto-buccal and mid-palatinal) and scores between 0- 3 were given for each point.
  Scoring was made as follows:
  0 - No microbial dental plaque in the gingival area
  1. - A film of microbial dental plaque adhering to the free gingival margin and adjacent area of the tooth, recognized only by running a probe across the tooth surfaces.
  2. - Moderate accumulation of soft deposits within the gingival pocket and on the gingival margin and/or adjacent tooth surfaces that can be seen by the naked eye.
  3. - Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.
Gingival Index | 12 months
  The periodontal probe was used to assess the bleeding potential of the tissues from 4 tooth surfaces (mesio-buccal papilla, mid-buccal margin, disto- buccal papilla and mid-palatinal margin) and scores between 0 - 3 were given for each point.
  Scoring was made as follows: 0 - Normal gingiva
  1. - Mild inflammation, slight change in color, slight edema; no bleeding on probing (BoP)
  2. - Moderate inflammation, redness, edema, and glazing; bleeding on probing
  3. - Severe inflammation, marked redness and edema, ulcerations; tendency to spontaneous bleeding.
Bleeding on Probing | 12 months
  The periodontal probe was used to assess the percentage of bleeding after probing from 4 tooth surfaces (mesio-buccal papilla, mid-buccal margin, disto-buccal papilla and mid-palatinal margin) and scored as positive (+) or negative (-) bleeding for each point.
Probing Depth | 12 months
  Probing Depth of the recession defect was measured in mm by the periodontal probe at the mid buccal surface of the related tooth as the distance between the gingival margin and the bottom of the gingival sulcus.
Clinical Attachment Level | 12 months
  Clinical Attachment Level of the recession defect was measured in mm by the periodontal probe at the mid-buccal surface of the related tooth and it was defined as the distance between the cemento-enamel junction and the bottom of the gingival sulcus
Recession Depth | 12 months
  Recession Depth was measured in mm by the periodontal probe at the mid-buccal surface of the related tooth as the distance between the cemento-enamel junction and the most apical point of the gingival margin
Recession Width | 12 months
  Recession Width of the defect was measured in mm by the periodontal probe as the horizontal distance from one border of the recession to another in mesio-distal direction at the level of the cemento-enamel junction
Gingival Thickness | 12 months
  Gingival Thickness was measured in mm at the mid-point location between the gingival margin and mucogingival junction, using an #25 endodontic spreader. Under the local anesthesia, the spreader was pierced perpendicularly to the mucosal surface, through the soft tissue with light pressure until hard surface was felt. The silicone disk stop was placed in tight contact with the external soft tissue surface. After carefully removing the spreader, penetration depth was measured with a digital caliper5 with 0.05 resolution.
Keratinized Tissue Width | 12 months
  Keratinized Tissue Width of the recession defect was measured in mm by the periodontal probe at the same point as the probing depth, clinical attachment level and recession depth.

CONTACTS AND LOCATIONS:
Overall Officials: Cavid Ahmedbeyli, PhD, Principal Investigator — Aziz Aliyev Azerbaijan State Advanced Training Institute for Doctors
Locations (4):
- Aziz Aliyev Azerbaijan State Advanced Training Institute for Doctors, Baku, Azerbaijan
- Ibirapuera University, São Paulo, Brazil
- El Bosque University, Bogotá, Colombia
- Altinbas University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No